CLINICAL TRIAL: NCT01316068
Title: Effect of Intravenous and Oral Therapy With Sulodexide on Albuminuria in Type 2 Diabetic Patients
Brief Title: Effect of Sulodexide on Albuminuria in Chinese Type 2 Diabetic Patients
Acronym: Soften
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Collaborators: ALFA WASSERMANN（BJ) Market Research and Management Co., Ltd (Unknown)
Responsible Party: endocrinology department of the first affiliated hospital of Sun Yat-sen University, Yanbing Li
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sulodexide20110311
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2010-08

CONDITIONS: Diabetic Nephropathy; Albuminuria
Keywords: diabetic nephropathy; albuminuria; type 2 diabetes; sulodexide
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequencial use of sulodexide (Experimental): Patients will be given sulodexide 1200 LSU per day intravenously for 2 weeks. Then patients will receive 1000 LSU per day orally for 50 weeks.
  Interventions: Drug: intravenous use of sulodexide followed by oral use
- oral use of sulodexide (Active Comparator): Patients allocated to oral group will received 1000 LSU per day orally for 52 weeks
  Interventions: Drug: use of sulodexide orally only

INTERVENTIONS:
Drug: intravenous use of sulodexide followed by oral use — Patients will be given sulodexide 1200 LSU per day intravenously for 2 weeks,then receive 1000 LSU per day orally for 50 weeks.
  Other Names: sequential use of sulodexide
  Arms: sequencial use of sulodexide
Drug: use of sulodexide orally only — Patients receive 1000 LSU per day orally for 52 weeks
  Other Names: oral use of sulodexide
  Arms: oral use of sulodexide

SUMMARY:
Current therapies targeting albuminuria in diabetic nephropathy leave residual urinary albumin secretion, which meanwhile leave residual cardiovascular risk. Previous studies demonstrated that sulodexide could reduce albuminuria in type 2 diabetic patients. But no data concerning Chinese population is available. The investigators aim to provide evidence of effects of sulodexide on diabetic nephropathy in Chinese diabetic patients. Further the investigators also test the hypothesis that sequential administration of intravenous and oral replacement of the drug would gain an earlier and greater reduction of albuminuria, compared with oral use only.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes based on WHO criteria
* Age 18-75 years old
* Serum creatinine ≤ 1.5 mg/dL (130umol/L)
* Albuminuria defined by a urine albumin/creatinine ratio(ACR) according to ADA criteria 2009 (microalbuminuria by 30-299 ug albumin/mg creatinine and macroalbuminuria by ≥300 ug albumin/mg creatinine on random spot urine collection )
* Continued stable seated systolic blood pressure < 180 mmHg and diastolic blood pressure < 110 mmHg
* Willing to change antihypertensive medication regimen if necessary
* Willing to provide written informed consent to participate in the study
* Willing to take contraception,or infertility for the duration of the study

Exclusion Criteria:

* Type 1 diabetes mellitus
* Present acute diabetic complication, or severe chronic diabetic complication(e.g. proliferative diabetic retinopathy)
* Complicating uncontrolled severe infection
* Hepatic insufficiency or renal insufficiency or severe disturbance of lipid metabolism
* Blood pressure ≥ 180/110mmHg
* Severe concomitant systemic disease(e.g. cardiac insufficiency, stroke), anticipated to be unable to finish the trial
* Uncooperative,unable to follow up, or anticipated unable to finish the trial
* Patients with other known specific renal diseases
* Untreated urinary tract infection that would impact urinary protein values
* Evidence of hepatic dysfunction including total bilirubin > 2.0 mg/dL (34 mmol/L) or elevated transaminases
* History of Cardiovascular disease as follows: Unstable angina pectoris, myocardial infarction, transient ischemic attack, cerebrovascular accident, New York Heart Association Functional Class III or IV heart failure, obstructive valvular heart disease or hypertrophic cardiomyopathy
* Any risk of bleeding, or platelet count < 100×109/L or anticipated surgery within research period
* Active, recurrent or metastatic cancer, or known HIV infection
* Participant in any experimental drug study in the past 90 days prior to the enrollment of the study, or plan to participate in any drug study during the study period
* Prior exposure to sulodexide, either in a clinical setting or as a participant in another clinical study
* Known allergy or intolerance to any heparin-like compounds or multiple drug allergies
* Lactation, pregnancy, or an anticipated or planned pregnancy during the study period
* Inability to give an informed consent or to cooperate with researchers (e.g. psychiatric disorder) or history of noncompliance to medical regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in urine albumin/creatinine ratio | 52th week since the commence of therapy
  conversion to normoalbuminuria and at least a 25% reduction in UACR opposed to baseline, or 50% reduction in UACR opposed to baseline

SECONDARY OUTCOMES:
Change from Baseline in urine albumin/creatinine ratio and serum creatinine | before and 2nd,12th,24th,36th and 60th week since the commence of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Li, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Blouza S, Dakhli S, Abid H, Aissaoui M, Ardhaoui I, Ben Abdallah N, Ben Brahim S, Ben Ghorbel I, Ben Salem N, Beji S, Chamakhi S, Derbel A, Derouiche F, Djait F, Doghri T, Fourti Y, Gharbi F, Jellouli K, Jellazi N, Kamoun K, Khedher A, Letaief A, Limam R, Mekaouer A, Miledi R, Nagati K, Naouar M, Sellem S, Tarzi H, Turki S, Zidi B, Achour A; DAVET (Diabetic Albuminuria Vessel Tunisia Study Investigators). Efficacy of low-dose oral sulodexide in the management of diabetic nephropathy. J Nephrol. 2010 Jul-Aug;23(4):415-24. PMID 20175052
- [Background] Chen S, Fang Z, Zhu Z, Deng A, Liu J, Zhang C. Protective effect of sulodexide on podocyte injury in adriamycin nephropathy rats. J Huazhong Univ Sci Technolog Med Sci. 2009 Dec;29(6):715-9. doi: 10.1007/s11596-009-0608-0. Epub 2009 Dec 29. PMID 20037813
- [Background] Rossini M, Naito T, Yang H, Freeman M, Donnert E, Ma LJ, Dunn SR, Sharma K, Fogo AB. Sulodexide ameliorates early but not late kidney disease in models of radiation nephropathy and diabetic nephropathy. Nephrol Dial Transplant. 2010 Jun;25(6):1803-10. doi: 10.1093/ndt/gfp724. Epub 2010 Jan 7. PMID 20061322
- [Background] Lewis EJ, Xu X. Abnormal glomerular permeability characteristics in diabetic nephropathy: implications for the therapeutic use of low-molecular weight heparin. Diabetes Care. 2008 Feb;31 Suppl 2:S202-7. doi: 10.2337/dc08-s251. PMID 18227486
- [Background] Weiss R, Niecestro R, Raz I. The role of sulodexide in the treatment of diabetic nephropathy. Drugs. 2007;67(18):2681-96. doi: 10.2165/00003495-200767180-00004. PMID 18062718
- [Background] Sulikowska B, Olejniczak H, Muszynska M, Odrowaz-Sypniewska G, Gaddi A, Savini C, Cicero AF, Laghi L, Manitius J. Effect of sulodexide on albuminuria, NAG excretion and glomerular filtration response to dopamine in diabetic patients. Am J Nephrol. 2006;26(6):621-8. doi: 10.1159/000098195. Epub 2006 Dec 21. PMID 17191008
- [Background] Achour A, Kacem M, Dibej K, Skhiri H, Bouraoui S, El May M. One year course of oral sulodexide in the management of diabetic nephropathy. J Nephrol. 2005 Sep-Oct;18(5):568-74. PMID 16299683
- [Background] Gambaro G, Kinalska I, Oksa A, Pont'uch P, Hertlova M, Olsovsky J, Manitius J, Fedele D, Czekalski S, Perusicova J, Skrha J, Taton J, Grzeszczak W, Crepaldi G. Oral sulodexide reduces albuminuria in microalbuminuric and macroalbuminuric type 1 and type 2 diabetic patients: the Di.N.A.S. randomized trial. J Am Soc Nephrol. 2002 Jun;13(6):1615-25. doi: 10.1097/01.asn.0000014254.87188.e5. PMID 12039991
- [Background] Poplawska A, Szelachowska M, Topolska J, Wysocka-Solowie B, Kinalska I. Effect of glycosaminoglycans on urinary albumin excretion in insulin-dependent diabetic patients with micro- or macroalbuminuria. Diabetes Res Clin Pract. 1997 Nov;38(2):109-14. doi: 10.1016/s0168-8227(97)00096-x. PMID 9483374